CLINICAL TRIAL: NCT05136521
Title: A Randomized, Two-way Cross-over Comparative Bioavailability Study of 300 mg Trazodone Hydrochloride Containing New Polymer vs. 300 mg Trazodone Hydrochloride Containing Contramid® Prolonged-release Tablets Under Fasting Conditions
Brief Title: Bioavailability Study of 300 mg Trazodone Hydrochloride (New Polymer) vs. 300 mg Trazodone Hydrochloride (Contramid® Prolonged-release Tablets) Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aziende Chimiche Riunite Angelini Francesco S.p.A (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 039(C/a)WO19390; CRO-PK-19-340 (Other: CROSS Research)
Record Dates: First submitted 2021-11-02; First posted 2021-11-29 (Actual); Last update posted 2021-11-29 (Actual); Status verified 2021-11

CONDITIONS: Healthy
Keywords: Bioavailability; Cross over; trazodone hydrochloride (HCl) (new polymer); Trittico®, 300 mg trazodone HCl; Bioequivalence; prolonged-release tablets; Contramid®,
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — Trazodone

STUDY DESIGN:
Intervention Model Description: The study is single dose, open-label, randomised, two-period, two-sequence, cross-over, bioavailability and bioequivalence study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 300 mg trazodone hydrochloride (HCl) prolonged-release tablets (new polymer) (Experimental): Subjects treated with 300 mg trazodone HCl prolonged-release tablets containing a new polymer,
  Interventions: Drug: Trazodone HCl - new polymer
- Trittico®, 300 mg trazodone HCl prolonged-release tablets (Contramid®) (Active Comparator): Subjects treated with Trittico®, 300 mg trazodone HCl prolonged-release tablets containing Contramid®
  Interventions: Drug: Trazodone HCl - Contramid®

INTERVENTIONS:
Drug: Trazodone HCl - new polymer — A single 300 mg dose of the test (T) and of the reference (R) products will be administered to the study subjects in two consecutive periods, according to a randomised 2-sequence cross-over design. A wash-out interval of at least 10 days will elapse between the two administrations. The two investigational products will be administered with 240 mL of still mineral water on day 1 of the two study periods, at 08:00±1 h after an overnight fasting.
  Arms: 300 mg trazodone hydrochloride (HCl) prolonged-release tablets (new polymer)
Drug: Trazodone HCl - Contramid® — A single 300 mg dose of the test (T) and of the reference (R) products will be administered to the study subjects in two consecutive periods, according to a randomised 2-sequence cross-over design. A wash-out interval of at least 10 days will elapse between the two administrations. The two investigational products will be administered with 240 mL of still mineral water on day 1 of the two study periods, at 08:00±1 h after an overnight fasting.
  Other Names: Trittico®
  Arms: Trittico®, 300 mg trazodone HCl prolonged-release tablets (Contramid®)

SUMMARY:
This study was designed to investigate the bioequivalence of the test and reference products when administered as single oral doses in two consecutive study periods, under fasting conditions.

DETAILED DESCRIPTION:
A single 300 mg dose of the test (T) and of the reference (R) products will be administered to the study subjects in two consecutive periods, according to a randomised 2-sequence cross-over design. A wash-out interval of at least 10 days will elapse between the two administrations. The two investigational products will be administered with 240 mL of still mineral water on day 1 of the two study periods, at 08:00±1 h after an overnight fasting.

To investigate the bioequivalence of the test and reference products when administered as single oral doses in two consecutive study periods, under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent: signed written informed consent before inclusion in the study
* Sex and Age: men and women, 18-45 years old inclusive
* Body Mass Index (BMI): 18.5-30 kg/m2 inclusive
* Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest in the sitting position
* Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the Investigator and to comply with the requirements of the entire study
* Contraception and fertility : men and women of child-bearing potential and with an active sexual life must be using at least one of the following reliable methods of contraception throughout the study:
* Hormonal oral, implantable, intrauterine device [IUD], transdermal, or injectable contraceptives for at least 2 months before the screening visit (women only)
* A non-hormonal intrauterine device or female condom with spermicide or contraceptive sponge with spermicide or diaphragm with spermicide or cervical cap with spermicide for at least 2 months before the screening visit (women only)
* A male sexual partner who agrees to use a male condom with spermicide (women only)
* A vasectomised partner (women only)
* A male condom with spermicide (men only)
* A sterile sexual partner Female participants of non-child-bearing potential or in post-menopausal status for at least 1 year will be admitted

Exclusion Criteria:

* Electrocardiogram (ECG): clinically significant abnormalities at 12-lead ECG in supine position
* QTc: QTcF>430 msec for men and QTcF>450 msec for women at screening
* Cardiac disorders: history of risk factors for torsade de pointes, such as heart failure, significant cardiac arrhythmias, significant cardiac conduction abnormalities, family history of long QT syndrome, cardiac hypertrophy, cardiomyopathy, chronic cardiac insufficiency
* Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
* Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
* Allergy: ascertained or presumptive hypersensitivity to the active principle and/or formulations' ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study
* Diseases: history of significant renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study
* Medications: medications, including over the counter (OTC) medications and herbal remedies and in particular concomitant intake of potentially hepatotoxic drugs or hepatic/gastric enzyme inducers (i.e. phenobarbital, phenytoin, carbamazepine, chlorzoxazone and rifampicin) for 2 weeks before the start of the study. Hormonal contraceptives for women will be allowed
* Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval will be calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
* Blood donation: blood donations for 3 months before this study
* Drug, alcohol, caffeine, tobacco: history of drug, alcohol [>1 drink/day for women and >2 drinks/day for men, defined according to USDA Dietary Guidelines 2015-2020 (18)], caffeine (>5 cups coffee/tea/day) or tobacco (> or equal 6 cigarettes/day) abuse;
* Drug test: positive drug test at screening or day -1
* Alcohol breath test: positive alcohol breath test at day -1
* Diet: abnormal diets (<1600 or >3500 kcal/day) or substantial changes in eating habits in the 4 weeks before this study; vegetarians
* Pregnancy: pregnant or lactating women; positive or missing pregnancy test at screening or day -1

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-07-19 (Actual); Study Completion 2020-07-19 (Actual)

PRIMARY OUTCOMES:
Cmax | At pre-dose (0) and 0.5, 1, 2, 3, 4, 5, 6, 8, 9, 10, 11, 12, 14, 16, 20, 24, 30, 36, 48, 72, 96 hours post-dose
  Cmax of plasma trazodone (free base). The following PK parameter will be measured and/or calculated for plasma trazodone (free base) applying a Non-Compartmental Analysis, using the validated software Phoenix WinNonlin® version 6.3 (22) or higher (the actual version will be stated in the final report).
AUC(0-t) | At pre-dose (0) and 0.5, 1, 2, 3, 4, 5, 6, 8, 9, 10, 11, 12, 14, 16, 20, 24, 30, 36, 48, 72, 96 hours post-dose
  AUC(0-t) of plasma trazodone (free base). The following PK parameter will be measured and/or calculated for plasma trazodone (free base) applying a Non-Compartmental Analysis, using the validated software Phoenix WinNonlin® version 6.3 (22) or higher (the actual version will be stated in the final report).
AUC(0-∞) | At pre-dose (0) and 0.5, 1, 2, 3, 4, 5, 6, 8, 9, 10, 11, 12, 14, 16, 20, 24, 30, 36, 48, 72, 96 hours post-dose
  AUC(0-∞) of plasma trazodone (free base). The following PK parameter will be measured and/or calculated for plasma trazodone (free base) applying a Non-Compartmental Analysis, using the validated software Phoenix WinNonlin® version 6.3 (22) or higher (the actual version will be stated in the final report).

SECONDARY OUTCOMES:
Treatment emergent adverse events (TEAEs) | Trough study completion, an average of five months
  All AEs occurring or worsening after the first dose of IMP. Adverse events (AEs) will be coded by System Organ Class (SOC) and Preferred Term (PT), using the Medical Dictionary for Regulatory Activities (MedDRA)
Residual area | At pre-dose (0) and 0.5, 1, 2, 3, 4, 5, 6, 8, 9, 10, 11, 12, 14, 16, 20, 24, 30, 36, 48, 72, 96 hours post-dose
  Residual area of plasma trazodone (free base). Extrapolated area calculated as (AUC(0-∞) - AUC(0-t))/ AUC(0-∞)
tmax | At pre-dose (0) and 0.5, 1, 2, 3, 4, 5, 6, 8, 9, 10, 11, 12, 14, 16, 20, 24, 30, 36, 48, 72, 96 hours post-dose
  Time to achieve Cmax of plasma trazodone (free base)
tlag | At pre-dose (0) and 0.5, 1, 2, 3, 4, 5, 6, 8, 9, 10, 11, 12, 14, 16, 20, 24, 30, 36, 48, 72, 96 hours post-dose
  Lag-time observed from the dosing time point prior to that of the first measurable plasma concentration (≥ LLOQ) (tlag ≥ 0) of plasma trazodone (free base)
λz | At pre-dose (0) and 0.5, 1, 2, 3, 4, 5, 6, 8, 9, 10, 11, 12, 14, 16, 20, 24, 30, 36, 48, 72, 96 hours post-dose
  λz is apparent terminal elimination rate constant, calculated, if feasible, by log-linear regression using at least 3 points of plasma trazodone (free base)
t1/2 | At pre-dose (0) and 0.5, 1, 2, 3, 4, 5, 6, 8, 9, 10, 11, 12, 14, 16, 20, 24, 30, 36, 48, 72, 96 hours post-dose
  Apparent terminal elimination half-life, calculated, if feasible, as ln2/λz,

CONTACTS AND LOCATIONS:
Locations (1):
- CROSS Research S.A., Phase I Unit, Via F.A. Giorgioli 14 Phone: Fax: +41.91.63.00.511 Email:, Arzo, Switzerland